CLINICAL TRIAL: NCT01164878
Title: Cholestasis in Extreme Low Birth Weight Infants (ELBW) - Possible Influences of a Change in Nutrition Policy
Brief Title: Cholestasis in Extreme Low Birth Weight Infants (ELBW)
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Nadja Haiden,MD, PD Dr., Medical University of Vienna
Other Study IDs: MUVNeo-1
Record Dates: First submitted 2010-07-12; First posted 2010-07-19 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Cholestasis
Keywords: Cholestasis; Liver damage; Parenteral Nutrition; Aggressive Nutrition; Preterm; Extreme low birth weight infant; Parenteral Nutrition Associated Cholestasis
MeSH Terms: conditions — Cholestasis; Hyperphagia; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Before: ELBW infants before change of feeding policy
- After: ELBW infants after change of feeding policy

SUMMARY:
Parenteral nutrition associated liver disease (PNALD) in preterm neonates is characterized by early occurrence of intrahepatic cholestasis (parenteral nutrition associated cholestasis (PNAC).

Extreme low birth weight infants (ELBW, birth weight < 1000 g) are at increased risk for development of PNAC.

Important factors implicated in the aetiology of PNAC are high caloric parenteral nutrition using amino acids or dextrose, but also intravenous lipids and infections in particular necrotizing enterocolitis (NEC).

Due to a change of paradigm a more aggressive nutrition with early use of parenteral amino acids/lipids and early fortification of mothers milk or alternatively high caloric preterm formula is warranted. Accordingly - in line with the existing expert opinion and evidence - the feeding policy at the neonatal care units of our hospital was adapted.

Evidence exists that PNAC might be caused by the use of high concentrations of amino acids and lipids in parenteral nutrition. Furthermore NEC is associated with high osmotic feeds. Therefore the incidence of PNAC might be increased directly and indirectly after introducing the new feeding policy.

The investigators therefore aim at retrospectively investigating the incidence of PNAC before and after introduction of a feeding policy of "aggressive nutrition" for ELBW infants.

ELIGIBILITY:
Inclusion Criteria:

* ELBW infants below 1000 Gram birth weight
* Born in house between January 2005 - December 2006 ("before") and July 2007- June 2009 ("after")

Exclusion Criteria:

* signs of cholestasis at birth
* Death or transfer before 28 Days of life
* Diseases associated with Cholestasis

Max Age: 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm Infants below 1000 Gram birth weight
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Cholestasis | Assessment of bilirubin levels at least every second week from birth (0 weeks) to discharge (i.e. up to an average of 12 weeks)
  Conjugated Bilirubin > 1.5 mg/dl at two measurements

SECONDARY OUTCOMES:
Growth | At study entry (after birth, 0 weeks) and discharge (i.e. at an average of 12 weeks)
  Body weight, head circumference and heel-crown length assessed at birth and at discharge from or transfer to another hospital

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Haiden, MD, Principal Investigator — Medical University Vienna; Andreas Repa, MD, Principal Investigator — Medical University Vienna

REFERENCES:
- [Background] Repa A, Lochmann R, Unterasinger L, Weber M, Berger A, Haiden N. Aggressive nutrition in extremely low birth weight infants: impact on parenteral nutrition associated cholestasis and growth. PeerJ. 2016 Sep 20;4:e2483. doi: 10.7717/peerj.2483. eCollection 2016. PMID 27688976
- See also: Open source article — https://peerj.com/articles/2483/
- Available data/document: Individual Participant Data Set — https://dfzljdn9uc3pi.cloudfront.net/2016/2483/1/SPSS_repa_et_al.sav — SPSS Data Set for Analysis